CLINICAL TRIAL: NCT05770349
Title: Association of Ultrastructural Characteristics of Mitochondria in Cardiomyocytes and Signs of Mitochondrial Dysfunction With the Clinical Course and Outcomes of Heart Failure
Brief Title: Ultrastructural Characteristics of Mitochondria in Cardiomyocytes in Heart Failure
Acronym: MITOCH-HF
Status: Recruiting | Type: Observational
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Collaborators: Russian Science Foundation (Other)
Responsible Party: Principal Investigator, Elena A. Kuzheleva, Senior Researcher, Tomsk National Research Medical Center of the Russian Academy of Sciences
Other Study IDs: 23-75-00009
Record Dates: First submitted 2023-02-21; First posted 2023-03-15 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure; Coronary Artery Disease
Keywords: Chronic heart failure; Mitochondrial function; Mitochondrial DNA; Electron microscopy; SPECT; Cytochrome C; CABG
MeSH Terms: conditions — Heart Failure; Coronary Artery Disease | interventions — Coronary Artery Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — fixed tissue, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: coronary artery bypass grafting — Coronary artery bypass grafting

SUMMARY:
According to modern concepts, mitochondrial dysfunction may be the fundamental basis for the development and progression of CHF, including in patients undergoing myocardial revascularization. The processes of mitochondrial fusion, division and mitophagy are aimed at maintaining cellular homeostasis. A change in the balance of these processes can lead to the accumulation of damaged organelles with impaired functions. In patients with CHF, dysfunctional mitochondria are characterized by size dispersion, crist disorganization, and localization changes relative to myofibrils.

At the same time, the topic of the influence of mitochondrial dysfunction on the prognosis and clinical course of CHF remains debatable today. Direct study of the structural and functional features of mitochondria in human cardiomyocytes is an extremely difficult task, and therefore, such studies are carried out extremely rarely and on very limited cohorts. In the planned study, due to the long time of the study material recruitment, the ultrastructure of mitochondria in a large cohort of patients, ranging from 45 to 60 people, will be studied.

The aim of this study is to study the association of mitochondrial dysfunction with the clinical course and outcomes of CHF of ischemic etiology, as well as to assess the degree of compliance of indirect criteria of mitochondrial dysfunction with direct ultrastructural characteristics of mitochondria in cardiomyocytes.

This single-center prospective cohort study will involve 45-60 patients. The patients will have biopsy samples taken from the right auricle, as well as blood collection and preservation and its derivatives. Electron microscopy of myocardial samples will be performed to assess the ultrastructure of mitochondria of cardiomyocytes. The results of a direct study of mitochondria will be compared with indirect signs of mitochondrial dysfunction: the registration of the phenomenon of increased leaching of radiopharmaceuticals from the myocardium, an increase in the number of copies of mitochondrial DNA and the concentration of cytochrome C in the blood, the affiliation of mitochondrial DNA to haplogroup K. The results obtained in each of the research tasks will have high scientific significance and publication potential.

DETAILED DESCRIPTION:
According to modern concepts, mitochondrial dysfunction may be the fundamental basis for the development and progression of CHF, including in patients undergoing myocardial revascularization. The processes of mitochondrial fusion, division and mitophagy are aimed at maintaining cellular homeostasis. A change in the balance of these processes can lead to the accumulation of damaged organelles with impaired functions. In patients with CHF, dysfunctional mitochondria are characterized by size dispersion, crist disorganization, and localization changes relative to myofibrils.

At the same time, the topic of the influence of mitochondrial dysfunction on the prognosis and clinical course of CHF remains debatable today. Direct study of the structural and functional features of mitochondria in human cardiomyocytes is an extremely difficult task, and therefore, such studies are carried out extremely rarely and on very limited cohorts. In the planned study, due to the long time of the study material recruitment, the ultrastructure of mitochondria in a large cohort of patients, ranging from 45 to 60 people, will be studied.

The aim of this study is to study the association of mitochondrial dysfunction with the clinical course and outcomes of CHF of ischemic etiology, as well as to assess the degree of compliance of indirect criteria of mitochondrial dysfunction with direct ultrastructural characteristics of mitochondria in cardiomyocytes.

This single-center prospective cohort study will involve 45-60 patients. The patients will have biopsy samples taken from the right auricle, as well as blood collection and preservation and its derivatives. Electron microscopy of myocardial samples will be performed to assess the ultrastructure of mitochondria of cardiomyocytes. The results of a direct study of mitochondria will be compared with indirect signs of mitochondrial dysfunction: the registration of the phenomenon of increased leaching of radiopharmaceuticals from the myocardium, an increase in the number of copies of mitochondrial DNA and the concentration of cytochrome C in the blood, the affiliation of mitochondrial DNA to haplogroup K. The results obtained in each of the research tasks will have high scientific significance and publication potential.

The results of the study will be obtained by solving the following tasks:

1. To investigate the clinical and prognostic significance of mitochondrial dysfunction, confirmed by direct and indirect methods of investigation, in patients with CHF with stenosing atherosclerosis of the coronary arteries who underwent surgical myocardial revascularization in the prospective cohort study;
2. To study ultrastructural characteristics of mitochondria of cardiomyocytes from the auricle of the right atrium using a transmission electron microscope JEM-1400 (JEOL, Japan) in patients with CHF with reduced or mildly reduced left ventricular ejection fraction (HFrEF, HFmrEF) and stenosing atherosclerosis of the coronary arteries;
3. To evaluate the features of the mitochondrial genome, in particular, to determine whether the mitochondrial DNA belongs to haplogroup K, which may be associated with impaired adaptation to hypoxia due to the negative effect of guanine replacement on adenine at position 9055 (G9055A) [Strauss K.A. et al. Severity of cardiomyopathy associated with adenine nucleotide translocator-1 deficiency correlates with mtDNA haplogroup. Proc Natl Acad Sci U S A. 2013 Feb 26;110(9):3453-8. doi: 10.1073/pnas.1300690110] and its relation to the prognosis of the disease and the ultrastructure of mitochondria according to electron microscopy;
4. To study the association of the number of copies of mitochondrial DNA in blood plasma with ultrastructural signs of mitochondrial dysfunction in CMC;
5. To evaluate the content of the biochemical marker of mitochondrial damage - cytochrome C in the blood serum of patients with CHF and to identify the correlation of its concentration with the severity of structural and functional changes in mitochondria;
6. To assess the significance of the phenomenon of enhanced leaching of the radiopharmaceutical Tc99-MIBI from the myocardium and to determine the degree of correlation of the rate of leaching of Tc99-MIBI with the ultrastructural state of mitochondria, as well as with the clinical course and prognosis of CHF;
7. Calculate statistical parameters (sensitivity, specificity, degree of concordance) for each of the indirect signs of mitochondrial dysfunction and their totality in the diagnosis of mitochondrial ultrastructure disorders according to electron microscopy data and prediction of the clinical course and outcomes of CHF in patients undergoing surgical myocardial revascularization.

Thus, it is planned to prove for the first time in the world the association of direct ultrastructural signs of mitochondrial dysfunction with the clinical course and outcomes of CHF in patients who underwent surgical myocardial revascularization. For the first time in the world, the degree of compliance of available indirect signs of mitochondrial dysfunction with the true ultrastructural state of mitochondria will be presented, with the inclusion of 45-60 patients in the study. Based on the results of the study, a parameter or a set of parameters will be proposed that will be most associated with the clinical course of the disease and the outcome in patients with CHF of ischemic etiology.

The results obtained will have high world-class scientific significance and importance, both for fundamental medical science and for the practical implementation of the results.

ELIGIBILITY:
Inclusion Criteria:

1. The presence of HFrEF or HFmrEF (EF of LV <50%)
2. Obstructive multivessel coronary atherosclerosis as an indication for cardiac surgical correction of coronary blood flow (coronary bypass surgery)
3. Signed informed consent to participate in the study, separate consents for biomaterial sampling and genetic research

Exclusion Criteria:

1. Refusal of revascularization or participation in the study
2. Additional cardiac surgery other than coronary bypass surgery (valves, aneurysm)
3. Oncological diseases in the active stage;
4. The presence of implanted devices (EX, AICD, CT);
5. Severe renal dysfunction (GFR <30 ml/min/1.73 m2);
6. Infiltrative heart diseases (sarcoidosis, amyloidosis, accumulation diseases);
7. Autoimmune diseases;
8. Acute infectious and exacerbations of chronic somatic diseases
9. Type 1 or type 2 diabetes mellitus
10. Contraindications to myocardial scintigraphy, cardiopulmonary stress test
11. Impossibility of prescribing optimal drug therapy after cardiac surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 45-60 patients will be included in the study (15-20 people each - in 2023, 2024 and 2025) who meet the stated inclusion and exclusion criteria. The signing of the informed consent will be carried out before the start of any research procedures, the patient will be explained in detail the protocol of the study and the scope of the diagnostic procedures carried out
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint (combined) | 12 months
  cardiovascular death + hospitalization for decompensated HF or the need for parenteral administration of a diuretic + acute ischemic events or repeated unplanned revascularization + unplanned impalement of cardiac implantable electronic devices

SECONDARY OUTCOMES:
Duration of hospitalization | 30 days
  number of days of hospitalization
Postoperative complications during hospitalization | 30 days
  Postoperative complications during hospitalization
Worsening of NYHA class | 12 months
  Worsening of NYHA class
Dynamics of Echo parameters: left ventricular ejection fraction | 12 months
  Dynamics of left ventricular ejection fraction
Dynamics of NTproBNP | 12 months
  Change in the concentration of NTproBNP
Maximum oxygen consumption by cardiorespiratory stress test (Schiller ergospirometry system) | 12 months
  Change in maximum oxygen consumption
Dynamics of scores for the indicator "Physical health" according to the SF-36 questionnaire | 12 months
  Change in the quality of life index up or down
Dynamics of scores for the indicator "Mental health" according to the SF-36 questionnaire | 12 months
  Change in the quality of life index up or down
Dynamics of the quality of life according to the Minnesota questionnaire | 12 months
  Change in the quality of life index up or down

CONTACTS AND LOCATIONS:
Overall Officials: Alla A Garganeeva, Ph.D., Principal Investigator — Cardiology Research Institute, Tomsk National Research Medical Center, Russian Academy of Sciences
Locations (1):
- Tomsk National Research Medical Center, Russian Academy of Sciences, Tomsk, Russia

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Derived] Garganeeva AA, Kuzheleva EA, Tukish OV, Vitt KN, Kondratiev MY, Syromyatnikova EE, Andreev SL, Arsenieva YA, Korepanov VA, Afanasiev SA. Acute Decompensated Heart Failure: Structural and Functional Changes in Mitochondria. Kardiologiia. 2024 Dec 24;64(12):12-18. doi: 10.18087/cardio.2024.12.n2737. English, Russian. PMID 39784128